CLINICAL TRIAL: NCT03471052
Title: Randomised Controlled Trial of Radiofrequency Ablation Versus a Sham Procedure for Symptomatic Cervical Inlet Patch
Brief Title: Radiofrequency Ablation vs Sham Procedure for Symptomatic Cervical Inlet Patch
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 216038
Record Dates: First submitted 2018-03-07; First posted 2018-03-20 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Barrett Esophagus
MeSH Terms: conditions — Barrett Esophagus | interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiofrequency ablation (RFA) (Experimental): Radiofrequency ablation (RFA)
  Interventions: Procedure: Radiofrequency ablation (RFA)
- Sham procedure (No Intervention): Endoscopy will be performed under conscious sedation and all BarrX RFA equipment will be set up in room. A sound recording of the BarrxTM RFA device will be played (a distinct bell sound that is emitted from the generator) during the procedure.

INTERVENTIONS:
Procedure: Radiofrequency ablation (RFA) — Ablation using the Barrx RFA System is a new technique for field ablation in the oesophagus. It has been used for eradication of diseased epithelium of all three subclasses of Barrett's oesophagus (non-dysplastic Intestinal metaplasia (IM), Low grade dysplasia (LGD) and High grade dysplasia (HGD). The BarrxTM RFA System uses ultra short pulse RF energy delivering 40Watts/cm2 power density and 12Joule/cm2 energy density, and affects the mucosa whilst preserving the submucosa.
  Clinical trials have suggested that it is safe and effective for treating non-dysplastic IM, LGD and HGD in Barrett's oesophagus . Long term data show the effect to be durable over 5 years.
  Arms: Radiofrequency ablation (RFA)

SUMMARY:
Inlet patch is a congenital condition of the upper oesophagus, consisting of stomach lining that is in the wrong place. It affects 5% of the population. Symptoms are a feeling of a ball in the back of the throat (called chronic globus sensation), cough and sore throat - these account for 4% of general practitioner (GP) referral to Ear Nose & Throat departments.

There is no recognised treatment. Drugs that reduce acid may help but do not block mucus production. Argon Plasma coagulation has been shown to be successful but limited to a few expert centres. The investigators have previously shown a device that uses radiofrequency energy to remove the patch to be highly effective in a ten patient pilot study, with 80% response rate that was durable over 1 year.

The purpose of this trial is to demonstrate the previous study was not due to placebo effect alone, with a sham controlled arm. Patients would then crossover to treatment at 6 months after sham. All males and non-pregnant females over 18 years old with previously diagnosed inlet patch causing symptoms of globus, with > 50% severity on a visual analogue score, are eligible.

DETAILED DESCRIPTION:
Inlet patch is a congenital anomaly of the upper oesophagus, consisting of stomach lining that is in an aberrant position. Prevalence is up to 10% on endoscopy studies and 5% on post mortem studies. There is thought to be a link with another condition of the lower oesophagus called Barrett's oesophagus, although there is limited evidence. Unlike Barrett's oesophagus, progression to cancer from an inlet patch is exceptionally rare.

The inlet patch can produce acid and mucus, and is associated with symptoms including sore throat, cough and hoarseness. One particular symptom, called globus pharyngeus (the feeling of a ball in the back of the throat) is often associated with an inlet patch.

There is no recognised treatment for symptomatic inlet patch. Anti-acid medications works for some but not all, which may in part be explained by the lack of acid producing cells in some inlet patches. Ablation of the inlet patch has been successful in small series using Argon Plasma Coagulation. This device is, however, associated with inter user variability and unpredictable depth of ablation. Radiofrequency ablation (RFA) using the BarrxTM System is a National Institute for Health and Clinical Excellence (NICE) and FDA approved device for treatment of abnormal oesophageal lining, which has shown to be successful in reversing Barrett's oesophagus to normal squamous lining. These devices are advantageous as the depth of ablation is controlled. The investigators have previously demonstrated, in a pilot study, that these devices are safe and effective for reversal of inlet patch to normal mucosa, with improvement in symptoms.

This study will use the BarrxTM system to treat patients with symptomatic inlet patch that is refractory to standard anti-acid medication, in a blinded sham controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptoms secondary to Inlet patch and globus score > 50 on Visual Analogue Scale (VAS)
2. Histological confirmation of presence of Inlet patch
3. Symptoms not responsive or partially responsive to (proton pump inhibitor) PPI therapy for > = 6 weeks
4. Males and non-pregnant females over the age of 18 years. Female patients who are pre-menopausal must practice a medically acceptable form of contraception.
5. Patients must sign an informed consent form.

Exclusion Criteria:

1. Patients in whom endoscopy is contraindicated.
2. No globus symptoms
3. Patients previously or currently treated for oesophageal dysplasia or cancer
4. Patients with eosinophilic oesophagitis
5. Patients with oesophageal varices
6. Previous radiotherapy
7. Patients who have undergone Hellers myotomy
8. Pregnant females.
9. People under the age of 18 years.
10. Evidence of major motility disorder on High resolution Manometry
11. Patients with pre-existing ENT disorders causing globus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-03-06 (Actual); Primary Completion 2021-01-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Reduction in globus symptoms | 6 months post ablation
  >50% reduction in globus as assessed by improvement in patient symptom scoring
Endoscopic eradication of inlet patch | Change from 6 months to 12 months post final ablation
  Eradication of inlet patch as assessed by endoscopic investigation
Histological reversal to squamous mucosa | Change at 6 and 12 months
  Complete histological reversal to squamous mucosa as assessed by histological staining of the biopsy samples
Change in surface area of residual inlet patch post ablation | Change at 6 and 12 months
  Change in surface area of residual inlet patch post ablation

SECONDARY OUTCOMES:
Oesophageal pH pre and post ablation | Change at Pre-screening and 12 months
  Oesophageal pH pre and post ablation
Adverse events | Through study completion, an average of 12 months
  Adverse event incidence at any time during the study
Presence of buried mucosa consistent with inlet patch | During endoscopy
  Presence of buried mucosa consistent with inlet patch
Symptomatic response for cough, hoarseness and sore throat using Visual Analogue Scale (VAS) | Through study completion, an average of 12 months
  Symptomatic response for cough, hoarseness and sore throat using VAS

CONTACTS AND LOCATIONS:
Overall Officials: Jason Dunn, Principal Investigator — Consultant Gastroenterology
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No